CLINICAL TRIAL: NCT04659629
Title: A First-in-Human Phase 1 Study of NL-201 Monotherapy and in Combination With Pembrolizumab in Patients With Relapsed or Refractory Cancer
Brief Title: NL-201 Monotherapy and in Combination With Pembrolizumab in Patients With Relapsed or Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogene Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL201-101
Record Dates: First submitted 2020-11-09; First posted 2020-12-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor; Advanced Solid Tumor
Keywords: Cancer; NL-201; NL201-101; Phase 1; Immunotherapy; Cytokine; Pembrolizumab; Keytruda; IL-2; IL-15; MK-3475
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: NL-201 Monotherapy Dose Escalation (Experimental): NL-201 given as monotherapy by intravenous administration testing ascending doses and two different schedules.
  Interventions: Drug: NL-201
- Part 2: NL201 Monotherapy Expansion Cohorts (Experimental): NL-201 given as monotherapy by intravenous administration in indication specific cohorts at a dose and schedule determined in Part 1.
  Interventions: Drug: NL-201
- Part 3: NL-201 in Combination with Pembrolizumab Dose Escalation (Experimental): NL-201, in combination with a set Pembrolizumab dose, testing ascending doses and two different schedules
  Interventions: Drug: NL-201; Drug: Pembrolizumab Injection [Keytruda]
- Part 4: NL-201 in Combination with Pembrolizumab Expansion Cohorts (Experimental): NL-201 in combination with Pembrolizumab in indication specific cohorts at a dose and schedule determined in Part 3
  Interventions: Drug: NL-201; Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Drug: NL-201 — NL-201 is a de novo protein therapeutic.
Drug: Pembrolizumab Injection [Keytruda] — A programmed death receptor-1 (PD-1)-blocking antibody
  Other Names: MK-3475, Pembrolizumab, Keytruda
  Arms: Part 3: NL-201 in Combination with Pembrolizumab Dose Escalation; Part 4: NL-201 in Combination with Pembrolizumab Expansion Cohorts

SUMMARY:
Parts 1 and 2 The primary purpose of this study is to understand the safety of NL-201 when given intravenously as monotherapy in patients with advanced cancer to evaluate tolerability and to identify a recommended dose and schedule for further testing. In Part 1, there will be backfill cohorts at certain Data Monitoring Committee (DMC)-cleared dose levels and schedules to collect pharmacokinetic (PK), pharmacodynamic (PD) and response data in certain tumor types or to explore additional pre-medication regimens.

Parts 3 and 4 The primary purpose of this study is to understand the safety of NL-201 in combination with pembrolizumab when both drugs are given intravenously in patients with advanced cancer, to evaluate tolerability, and to identify a recommended dose and schedule for further testing.

DETAILED DESCRIPTION:
Patients will have tests and exams to see if they are eligible for the clinical trial.

Parts 1 and 2 If eligible, the patient will receive NL-201 treatment by vein. Tumor response to treatment will be assessed every 6 weeks for 12 weeks, and every 12 weeks thereafter until disease progression.

Patients will be able to receive study treatment as long as it is tolerated and there is evidence of clinical benefit. Safety follow-up will occur within 7 days after the last dose of NL-201. Patients will then enter long-term follow-up until starting a subsequent therapy.

In Part 1, there will be backfill cohorts at certain DMC-cleared dose levels and schedules to collect PK, PD and response data in certain tumor types or to explore additional pre-medication regimens.

Parts 3 and 4 If eligible, the patient will receive NL-201 and pembrolizumab treatment by vein. Tumor response to treatment will be assessed every 6 weeks for 12 weeks, and every 12 weeks thereafter until disease progression.

Patients will be able to receive study treatments as long as they are tolerated and there is evidence of clinical benefit. Safety follow-up will occur within 7 days after the last dose of investigational product. Patients will then enter long-term follow-up until starting a subsequent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable disease
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least 6 weeks from any prior nitrosurea or mitomycin C therapy; at least 4 weeks from any other prior chemotherapy or checkpoint inhibitor; at least 2 weeks from any kinase inhibitor
* Part 1 Only: Patients with relapsed or refractory advanced solid tumor, other than prostate cancer, who have progressed, not tolerated or are ineligible for all approved lines of therapy
* Part 2 Only: Patients with kidney and skin cancer who have failed at least 1 line of systemic therapy
* Part 3 Only: Patients with solid tumors who have received ≥ 1 prior line of therapy for advanced or metastatic disease
* Part 4 Only: Patients with diagnosed target disease OR previously received pembrolizumab

Exclusion Criteria:

* Prostate Cancer
* Any serious medical condition or laboratory abnormality or psychiatric condition or any other significant or unstable concurrent medical illness (in the opinion of the Investigator) would preclude protocol adherence or would make the safety of the study drug difficult to assess
* Known or suspected SARS-CoV-2 infection, unless patient tests negative for SARS-CoV-2 within the Screening period
* History of solid organ transplant or bone marrow transplant
* Prior chimeric antigen receptor T-cell (CAR-T) or allogeneic cellular therapy
* Prior IL-2-based cancer therapy
* Ongoing systemic immunosuppressive therapy
* Concurrent therapy with any other investigational agent, vaccine, or device.
* Part 3 and 4 Only: History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Part 3 and 4 Only: Known additional cancer that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone curative resection are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) for NL-201 (Parts 1 and 2) | Up to Day 33
  Evaluation of tolerability of NL-201 as measured by number of subjects with dose limiting toxicities (DLTs)
Recommended dose schedule for NL-201 (Parts 1 and 2) | Up to Day 33
  Evaluation of tolerability of NL-201 as measured by number of subjects with dose limiting toxicities (DLTs)
Recommended phase 2 dose (RP2D) for NL-201 in combination with Pembrolizumab (Parts 3 and 4) | Up to Day 33
  Evaluation of tolerability of NL-201 in combination with Pembrolizumab as measured by number of subjects with dose limiting toxicities (DLTs)
Recommended dose schedule for NL-201 in combination with Pembrolizumab (Parts 3 and 4) | Up to Day 33
  Evaluation of tolerability of NL-201 in combination with Pembrolizumab as measured by number of subjects with dose limiting toxicities (DLTs)
Incidence of treatment-emergent adverse events | Up to Day 33
  Rate of adverse events in patients with advanced solid tumors
Severity of treatment-emergent adverse events | Up to Day 33
  Rate of adverse event grades in patients with advanced solid tumors

SECONDARY OUTCOMES:
Best Objective Response according to RECIST version 1.1 | Up to 36 months
  Based on Investigator assessment of radiographic imaging
Objective Response Rate (ORR) according to RECIST version 1.1 | Up to 36 months
  Based on Investigator assessment of radiographic imaging
Progression-Free Survival (PFS) according to RECIST version 1.1 | Up to 36 months
  Based on Investigator assessment of radiographic imaging
Duration of Response (DOR) according to RECIST version 1.1 | Upto 36 months
  Based on Investigator assessment of radiographic imaging
Pharmacokinetic (PK) profile of NL-201 by half-life (t1/2) | Up to 24 Months
  Prespecified timepoints in serum before and after dosing with NL-201.
Pharmacokinetic (PK) profile of NL-201 by area under the plasma concentration time curve (AUC) | Up to 24 months
  Prespecified timepoints in serum before and after dosing with NL-201.
Pharmacokinetic (PK) profile of NL-201 by maximum observed plasma concentration (Cmax) | Up to 24 months
  Prespecified timepoints in serum before and after dosing with NL-201.
Pharmacokinetic (PK) profile of NL-201 by volume of distribution (Vd) | Up to 24 Months
  Prespecified timepoints in serum before and after dosing with NL-201.
Terminal-Phase Elimination Rate Constant (β) of NL-201 | Up to 24 months
  Prespecified timepoints in serum before and after dosing with NL-201.
Immunogenicity of NL-201 | Up to 24 months
  Anti-drug antibodies in serum during and after treatment with NL-201

OTHER OUTCOMES:
Flow cytometry analysis of immune cells in blood | Up to 36 months
  Based on appropriate assay
Serum measurements of inflammatory cytokine levels | Up to 36 months
  Based on appropriate assay
Analysis of immune characteristics of the tumor microenvironment | Up to 36 months
  Based on appropriate assay
Estimate additional measures of anti-tumor activity of NL- 201 per iRECIST criteria | Up to 36 months
  Based on Investigator assessment of imaging

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni A Razak, Principal Investigator — UHN - Princess Margaret Cancer Center
Locations (8):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Cancer Center Oncology and Hematology Care Clinic, Portland, Oregon
  - UT- MD Anderson, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - Melanoma Institute Australia, Sydney, New South Wales
  - St Vincents Hospital, Sydney, New South Wales
  - Olivia Newton-John Cancer Wellness & Research Centre, Heidelberg, Victoria
- UHN - Princess Margaret Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT04659629/Prot_SAP_000.pdf